CLINICAL TRIAL: NCT00957294
Title: The Metabolic Syndrome in Patients With First-episode Schizophrenia - Prognosis and Prediction.
Brief Title: Metabolic Syndrome in Patients With First-episode Schizophrenia
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Other Study IDs: Lene Nyboe Jacobsen
Record Dates: First submitted 2009-08-03; First posted 2009-08-12 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2012-03

CONDITIONS: Metabolic Syndrome X; Schizophrenia
MeSH Terms: conditions — Metabolic Syndrome; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Schizophrenia: Patients with first-episode schizophrenia age 18-45 years
- Depression: First-time hospitalized patients with depression age 18-45 years
- healthy controls: Healthy controls matched on age and gender (18-45 years)

SUMMARY:
The metabolic syndrome (MetS) is highly prevalent in patients with schizophrenia and is a major risk factor of type-2 diabetes, cardiovascular disease and early death. Genetic factors, antipsychotic medication, sleeping disturbances and unhealthy lifestyle are possible causes of developing metabolic syndrome. Several studies have investigated the metabolic side-effects of antipsychotic medication. However it is still unanswered how unhealthy lifestyle, comprising physical inactivity, smoking, unhealthy dieting, and sleeping disturbances adds to the metabolic risk of patients with schizophrenia. The aim of this study is to investigate the prevalence and development of MetS in first-episode patients with schizophrenia and 1 year after onset of treatment. The study's main hypothesis is that physical inactivity, regardless of medication, is an independent risk factor for metabolic syndrome in patients with schizophrenia. In comparison inpatients with major depression and healthy controls, both matched on gender, age and level of education will be included in the study. It is anticipated that the study's results will provide new knowledge about the risk of developing metabolic syndrome in first-episode schizophrenia and how different risk factors contribute to this.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ICD-10 diagnosed schizophrenia

Exclusion Criteria:

* Antipsychotic medication > 6 weeks before inclusion
* Physical disability
* Pregnancy
* IQ< 55

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients admitted to The OPUS project, Region of Midtjylland, Denamrk In comparison in-patients with major depression, Aarhus University Hospital, Risskov and healthy controls matched on gender, age and level of education.
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2009-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
metabolic syndrome | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Research Unit, Dep. Q of Affective Disorders, Aarhus University Hospital, Risskov, Aarhus, Risskov, Denmark